CLINICAL TRIAL: NCT02128412
Title: Expansion of Intracoronary Stents by Low Pressure Oversizing Versus High Pressure Inflation: A Randomised Intracoronary Ultrasound Controlled Study
Brief Title: IVUS Controlled Stenting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sydney South West Area Health Service (Other Government)
Responsible Party: Principal Investigator, Esther Zhou, Research Medical Student, Sydney South West Area Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/167
Record Dates: First submitted 2014-04-28; First posted 2014-05-01 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Angioplasty and Stenting; Single de Novo Coronary Artery Stenoses
Keywords: Patients scheduled to undergo coronary angioplasty and stenting because of symptoms related to a single de novo coronary artery stenoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stent oversize group (Active Comparator): Oversized stent deployed at low pressure:
  A stent premounted on a balloon with a nominal diameter halfway between the lumen diameter and the true vessel diameter (approximated by external elastic lamina) as assessed by IVUS. This will be based on the smallest of the vessel reference diameters proximal and distal to the lesion. In addition the vessel diameter must be greater than this diameter throughout the length of the lesion. This stent will be implanted at an inflation pressure of 10 atmospheres or less for at least 15 seconds and a second IVUS will be performed to assess the end point.
  Interventions: Device: Oversized stent deployed at low pressure (Multi-Link Bare Metal Stent or Xience Prime Evenolimus Eluting Stent)
- High pressure group (Active Comparator): Stent deployed at high pressure:
  A stent premounted on a balloon with a nominal diameter approximately equal to the vessel segment lumen reference diameter as previously assessed by IVUS will be used. This stent will be implanted at an inflation pressure of 14 atmospheres or more for at least 15 seconds and a second IVUS will be performed to assess the end point
  Interventions: Device: Stent deployed at high pressure (Multi-Link Bare Metal Stent or Xience Prime Evenolimus Eluting Stent)

INTERVENTIONS:
Device: Oversized stent deployed at low pressure (Multi-Link Bare Metal Stent or Xience Prime Evenolimus Eluting Stent) — Stent can include both bare metal stents and drug eluting stents. Depending on availabilities, different stent brands may be used.
  Arms: Stent oversize group
Device: Stent deployed at high pressure (Multi-Link Bare Metal Stent or Xience Prime Evenolimus Eluting Stent) — Stent can include both bare metal stents and drug eluting stents. Depending on availabilities, different stent brands may be used.
  Arms: High pressure group

SUMMARY:
Stent placement is now widely accepted to improve the results of angioplasty (an operation to widen the blood vessel) and decreasing the need for further surgery. Despite their worldwide acceptance, stent usage is still limited by renarrowing which occurs within the stent (restenosis) in some patients within the first six months. In addition there still exists a small risk of heart attacks soon after the stent is placed.

The purpose of this study is to test the safety and tolerability of trying to place the stents using a different strategy of using low pressure oversized balloon inflations as opposed to the usual high pressure balloon inflations. This may reduce injury to the artery and reduce the chance of renarrowing of the stent. In order to ensure this is a safe and effective way of performing the procedure the investigators intend to use an Intravascular ultrasound (IVUS) catheter to look from inside the artery at the stents. IVUS has proven to be the best way of ensuring optimal stent placement.

Primary hypothesis: Stents will be equally well expanded and apposed using a strategy of oversized stenting at normal inflation pressures ( < 10 atmospheres ) as compared to high pressure inflation (≥14 atmospheres) as guided by intravascular ultrasound imaging.

Secondary Hypothesis: There will be no difference in acute clinical endpoints (death, myocardial infarction, urgent revascularisation or stent thrombosis) using a strategy of oversized stenting at normal inflation pressure as compared to high pressure inflation.

Tertiary Hypothesis: If the above is shown to be true the investigators would hope to expand the study in order to reveal a decrease in stent restenosis using a strategy of lower pressure balloon inflations. The investigators will assess the deployment characteristics of drug eluting versus bare metal stents

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for a coronary angioplasty and stenting
* Single de novo artery stenosis are eligible for this study
* Target lesion needs to be less than 30mm long and located in a vessel more than 2.5 mm in diameter

Exclusion Criteria:

* Contraindication to antiplatelet therapy;
* Ostial lesion;
* Excessive vessel tortuosity;
* Lesion at a significant bifurcation (subbranch ≥ 2mm in diameter);
* Suspected intracoronary thrombus.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Number of stents which are optimally deployed as assessed against the MUSIC criteria | Immediately after stent is deployed until optimal deployment is achieved
  The criteria for optimal stent expansion are:
  1. Complete apposition of the stent over its entire length against the vessel wall.
  2a. In stent minimal luminal area (MLA) >= 90% of the average reference luminal area or >=100% of lumen area of the reference segment with the lowest lumen area.
  In stent lumen area of proximal stent entrance >= 90% of proximal lumen area. 2b. Where the instent luminal area is in excess of 9.0 mm2 , the following criteria apply: In stent MLA > 80% of the average reference lumen area or >=90% of lumen area of the reference segment with the lowest lumen area.
  In stent lumen area of proximal stent entrance >= 90% of proximal lumen area. 3. Symmetric stent expansion defined by lumen diameter (LD)min / LD max >= 0.7
  A less rigorous criteria for stent expansion will also be assessed:
  1. In stent MLA > 80% of the average reference lumen area; &
  2. Complete apposition of the stent over its entire length against the vessel wall

SECONDARY OUTCOMES:
Clinical endpoints including death, myocardial infarction, coronary artery bypass surgery, repeat percutaneous intervention, stent thrombosis, myonecrosis | 1-3 days following procedure and at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Craig Juergens, Cardiologist, Principal Investigator — South West Sydney, Liverpool
Locations (1):
- Department of Cardiology, Liverpool, New South Wales, Australia